CLINICAL TRIAL: NCT03053037
Title: Impact of Final Apical Size Preparation on Root Canal Treatment Success: A Clinical, Microbiological and Volumetric Evaluation
Brief Title: Apical Size and Root Canal Treatment Success Trial (AS-RCT Trial)
Acronym: AS-RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: American Association of Endodontists (Other)
Responsible Party: Principal Investigator, Vanessa Chrepa DDS, MS, Assistant Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 51641
Record Dates: First submitted 2017-02-10; First posted 2017-02-14 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Root Canal Therapy
Keywords: apical size; root canal treatment success; micro biome analysis; pulp necrosis
MeSH Terms: conditions — Dental Pulp Necrosis

STUDY DESIGN:
Intervention Model Description: randomized clinical trial 2 arms
Who Masked: Participant, Outcomes Assessor
Masking Description: Similar instrumentation method is used for both groups, therefore participants cannot be aware of the allocation. Data will be de-identified prior to outcome assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group S (Active Comparator): mesial canals in Group S will be instrumented to size 25
  Interventions: Procedure: final apical size instrumentation
- Group L (Active Comparator): mesial canals in Group L will be instrumented to size 35
  Interventions: Procedure: final apical size instrumentation

INTERVENTIONS:
Procedure: final apical size instrumentation — root canal instrumentation to two different final preparation sizes

SUMMARY:
This study is looking into two different ways to perform a root canal treatment. The study will look at differences and compare the two different treatment options over a 2-year period.More specifically, this study evaluates a small "skinny" root canal shape compared to a larger "broad" root canal shape and if this affects the success of the root canal treatment. Both types of treatment are standard of care and aim to treat the infection inside your tooth. When a tooth is infected with bacteria, we can see a dark area on the radiograph around the roots of the infected tooth. If this dark area becomes smaller or goes away completely after root canal treatment and you do not feel any pain or other symptoms, then we know that the treatment was successful and there is no need for further treatment on this tooth. To measure the size of the dark area around the tooth (i.e. volume) before and after the treatment we will need to take two limited volume three-dimensional radiographs (cone beam computed tomography-CBCT), one prior to treatment and one at two years after the root canal treatment is completed. These radiographs are more accurate in detecting changes in lesion size than the regular periapical radiographs. We will assess the changes in lesion volume for all teeth included in the study and that will help us find differences in success between the two root canal treatment protocols, We are specifically looking for persons that have been diagnosed with a necrotic permanent mandibular molar with an evident radiographic lesion (i.e. dark area around the tooth) that can be retained in the mouth with root canal treatment and permanent restoration. This study place participants in different treatment groups after randomization. Randomization means that you are placed by chance (like flipping a coin) into a treatment group. For this study, there are two treatment groups (protocol) and they are listed below.

Protocol 1: Group S: Root canal treatment will be performed in 2-visits using hand files and rotary instruments to a final canal shape of size #25.

Protocol 2: Group L: Root canal treatment will be performed in 2-visits using hand files and rotary instruments to a final canal shape of size #35

DETAILED DESCRIPTION:
We will perform a randomized, blinded clinical trial with clinical, microbiological and volumetric outcomes. The study population will be selected from adult patients in need of endodontic treatment on mandibular molars diagnosed with pulp necrosis and presenting with a visible radiographic lesion associated with at least the mesial root. Patients will be randomized into one of the two arms (group S: apical size#25; group L: apical size#35) and followed for 2 years post-treatment.

Treatment sequence Endodontic residents under the direct supervision of a study investigator will perform all treatments; all providers will be trained and calibrated for root canal treatment protocol and microbial sample collection. The calibration session will be repeated annually until completion of the study.

Treatment protocol First Appointment

1. Pre-operative CBCT will be obtained and baseline clinical signs and symptoms will be recorded. Pain level will be recorded on a 0-10 visual analog scale (VAS).
2. After ascertaining adequate local anesthesia, rubber dam isolation will be obtained and the field will be disinfected with 3% hydrogen peroxide and 2.5% sodium hypochlorite (NaOCl) solution as previously described (37).
3. Access will be performed and the operative field will be again disinfected with 2.5% NaOCl followed by 5% sodium thiosulphate. A microbiological sample (S0) of the field will be obtained with paper points. S0 will be used as a negative control (i.e. sterility sample).
4. The mesial canal walls will then be touched lightly with hand files to disrupt bacterial biofilms and a microbiological specimen (S1) will be obtained (described in detail below).
5. Orifice will be enlarged with a Protaper Universal SX rotary file (Dentsply, Tulsa, OK) Apical patency will be determined with a size #10 hand file and working length will be obtained with the use of Root ZX apex locator (J Morita USA, Irving, CA) and verified with a PA radiograph.
6. Coronal 2/3 of mesial canal WL will be instrumented with Vortex Blue rotary file 25/06 (Dentsply). First apical binding file (FABF) will be recorded at this stage to serve as a covariable in the analyses.
7. Apical 1/3 instrumentation of mesial canals will be carried out according to assigned group as follows:

1. Group S: Instrumentation technique to working length (WL) using the sequence 15/04 →20/04 →25/04 →25/06 Vortex Blue rotary file system (Dentsply).

2. Group L: Instrumentation technique to WL using the sequence 15/04 →20/04 →25/04 →25/06 → 30/04 →35/04 Vortex Blue rotary file system (Dentsply).

8. Distal(s) canal instrumentation will be standardized for both groups as follows:

1. Coronal 2/3 of distal canal will be instrumented with Vortex Blue rotary file 25/06 2. Apical instrumentation to WL using the sequence 15/04 →20/04 →25/04 →25/06 → 30/04 →35/04→40/04 Vortex Blue rotary file system (Dentsply) 9. The canals will be irrigated using a 30-gauge side-vented needle with 6% NaOCl (10ml/canal) followed by 17% ethylenediaminetetraacetic acid (EDTA; 5ml/canal) followed by a final rinse of 6% NaOCl (10ml/canal) and 5% sodium thiosulfate (2ml/canal).

10. A microbiological specimen (S2) will be obtained from mesial canals, and then the canals will be dried with paper points.

11. Calcium hydroxide [Ca(OH)2] will be placed as an interim intracanal medicament and a temporary restoration consisted of Fuji II LC (GC Corp, Tokyo, Japan) will be placed in the access. A post-op radiograph will be made.

Second appointment (within 10-14 days)

1. Clinical signs and symptoms will be recorded. Pain level will be recorded on a VAS.
2. After ascertaining adequate local anesthesia, rubber dam isolation will be obtained and the field will be disinfected as described above.
3. Root canal system will be accessed and a second sterility microbiological sample will be obtained (S00).
4. Ca(OH)2 will be removed by irrigating with 6% NaOCl (10ml/canal) followed by 17% EDTA (5ml/canal) and a final rinse of 6% NaOCl (10ml/canal). This will be followed by irrigation with 5% sodium thiosulfate (2ml/canal).
5. A microbiological specimen (S3) will be obtained from mesial canals, and then the canals will be dried with paper points.
6. Final obturation will be performed with gutta-percha and AH+ sealer utilizing the continuous wave condensation technique.
7. Access will be restored permanently and patient will be referred to their dentist for full coverage restoration. Adequate existing full coverage restorations will remain in place. A post-op radiograph will be made.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults 18-85 years old, ASA I, II
* Mandibular molars with diagnosis of necrotic pulp and periapical lesion associated with at least the mesial root
* Lesion with Periapical Index score > 2 and largest lesion dimension <10mm
* Fully developed apices and patent root canals, good periodontal health (probing depth < 4mm)
* Confirmed restorability with crown restoration after root canal treatment or adequate existing full cuspal coverage restoration

Exclusion Criteria:

* ASA Class III or IV, immune-compromised patients, pregnant women, history of diabetes or bisphosphonate treatment
* Teeth with coronal cracks that extend below the CEJ, or with non-odontogenic periapical pathology and/or with not fully developed apices
* Molars with c-shape anatomy or middle medial canal
* Patients unable to present for a recall at one-year and/or two-year post-treatment or unwilling to participate

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2016-08-05 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-02-07 (Actual)

PRIMARY OUTCOMES:
Success of root canal therapy | 2 years
  Volumetric assessment of the periapical lesion between baseline and endpoint assessment

SECONDARY OUTCOMES:
Relationship between the number and taxa of bacteria remaining in the root canal at the time of obturation and treatment success between the two groups. | 2 years
  Culture-independent, molecular methods will be performed to quantify the total bacterial count before and after treatment in each group as well as identify the specific oral taxa in the root canal and their association to treatment success.

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Chrepa, DDS, MS, Principal Investigator — University of Washington
Locations (2):
- United States (2):
  - University of Texas Health Science Center, San Antonio, Texas
  - University of Washington Dental School, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No